CLINICAL TRIAL: NCT02516462
Title: In Vitro Maturation of Human Eggs
Acronym: IVM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Foundation for Fertility Research (Other)
Collaborators: Fertility Laboratories Of Colorado (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFFR-IVM-2015
Record Dates: First submitted 2015-07-30; First posted 2015-08-06 (Estimated); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Infertility; Reproductive Techniques, Assisted
MeSH Terms: conditions — Infertility; Helping Behavior | interventions — Follicle Stimulating Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IVM (Experimental): Immature oocytes recovered from each subject will be placed into IVM media for maturation.
  Interventions: Device: IVM media; Drug: Follicle Stimulating Hormone (FSH)

INTERVENTIONS:
Device: IVM media — Media to support the nuclear maturation and cytoplasmic competence of human oocytes in culture.
Drug: Follicle Stimulating Hormone (FSH) — Low dose FSH is administered to stimulate follicle growth.

SUMMARY:
Because a large proportion of the embryo's quality is dependent upon the egg, this investigation focuses on treatment of the oocyte during in vitro maturation (IVM). In typical IVF cycles, the egg is recovered when it is mature and ready to be fertilized. However, at this point the oocyte's quality has been set, and cannot be altered. Therefore, to have an impact on oocyte quality the use of in IVM is critical. Development of a successful IVM protocol for clinical use would not only provide an option for women of advanced maternal age, it would also reduce the cost of IVF due to fewer exogenous gonadotropins used for stimulation, and significantly lessen the risk of ovarian hyper-stimulation.

The objective of this research study is to evaluate a newly developed oocyte maturation media system for human clinical use in assisted reproductive technology (ART).

DETAILED DESCRIPTION:
The novel device (IVM media system), is designed to support nuclear maturation of immature oocytes recovered after minimal ovarian stimulation with no LH/hCG administration, and improve oocyte competence. This may result in development of a greater number of embryos to the blastocyst stage.

FSH is administered starting on cycle day 3 to stimulate follicle growth. When the leading follicle reaches 12-14 mm, egg retrieval will be scheduled. No hCG/LH trigger will be administered. Specially designed maturation media is used to collect and culture the immature eggs once recovered from the follicle. Once the eggs have matured in vitro, fertilization and embryo culture, vitrification and comprehensive chromosomal screening will be completed as per standard operating procedures.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women who desire to conceive and come to CCRM for infertility treatment using IVF will be candidates for this study.
* Women with PCOS
* Patients can be of any race, culture, sexual orientation or ethnicity.

Exclusion Criteria:

* Minors are excluded from participation in this study.
* Women with a BMI greater than 40
* Women whose health is such that becoming pregnant carries risk significantly greater than healthy women are excluded from this study, unless they use a gestational carrier under the direction of their physician.

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-07; Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Pregnancy | 6 months after egg retrieval
  The incidence of pregnancy following embryo transfer of IVM produced embryos.

SECONDARY OUTCOMES:
Development of good quality blastocysts using the Gardner morphological blastocyst grading system | 7 days after egg retrieval
  The proportion of good quality blastocyst stage embryos developed from IVM eggs during in vitro fertilization (IVF), of the total number of oocytes recovered
Offspring Weight | 1 year after egg retrieval
  The birth weight of children born following IVM
Offspring Gender | 1 year after egg retrieval
  The gender of children born after IVM
Fertilization of eggs | 2 days after egg retrieval
  The percentage of mature eggs that are successfully fertilized following IVM and IVF
Euploid Embryos | 1 month after egg retrieval
  The percentage of euploid embryos produced as analyzed by comprehensive chromosome screening, of total embryos tested

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca L Krisher, PhD, Study Director — CCRM
Locations (2):
- United States (2):
  - Fertility Laboratories of Colorado, Lone Tree, Colorado
  - National Foundation for Fertility Research, Lone Tree, Colorado